CLINICAL TRIAL: NCT02556736
Title: Phase I/IIa, Open-Label, Dose-Escalation Study of Safety and Tolerability of Intravitreal RST-001 in Patients With Advanced Retinitis Pigmentosa (RP)
Brief Title: AGN-151597 (Formerly RST-001) Phase I/II Trial for Advanced Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RST-001-CP-0001
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Retinitis Pigmentosa
Keywords: Gene therapy; Optogenetics; Channelrhodopsin; Retina; Retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1: Low Dose (Experimental): Single intravitreal injection of AGN-151597
  Interventions: Drug: AGN-151597
- Phase 1: Mid Dose (Experimental): Single intravitreal injection of AGN-151597
  Interventions: Drug: AGN-151597
- Phase 1: High Dose (Experimental): Single intravitreal injection of AGN-151597
  Interventions: Drug: AGN-151597
- Phase 2: High Dose (Experimental): Single intravitreal injection of AGN-151597
  Interventions: Drug: AGN-151597

INTERVENTIONS:
Drug: AGN-151597 — AGN-151597 is a gene therapeutic delivered by intravitreal injection

SUMMARY:
All participants in phase 1 and phase 2a had hand motion visual acuity or worse.

If efficacy was demonstrated from phase 1, better vision subjects could be enrolled; however, efficacy was not demonstrated.

DETAILED DESCRIPTION:
Study RST-001-CP-0001 was an open-label, dose-escalation study to evaluate the safety and tolerability of AGN-151597 (formerly RST-001) administered as a single intravitreal injection in participants with advanced RP. Three groups of approximately 3 participants each were sequentially enrolled in the dose-escalation phase (Phase 1) of this study: Group A (low dose), Group B (mid dose), and Group C (high dose).

For each dose group, the safety and tolerability of AGN-151597 was assessed by a data safety monitoring committee (DSMC) in the first participant before the remaining participants were enrolled into the group. If the DSMC considered the safety and tolerability of all participants in the dose group to be satisfactory and enrollment stopping rules had not been met, then enrollment into the next dose group could begin.

If the DSMC considered the safety and tolerability satisfactory and the enrollment stopping rules had not been met after a minimum assessment of 1 month (to include the Month 1 Visit) from treatment of the final participant in Groups A, B, or C, then the sponsor could elect to start enrollment of up to approximately 12 participants in Phase 2a to receive AGN-151597 at the maximum tolerated dose. After completion of the 2-year core study visits, each participant could enroll in a long-term follow-up for an additional 3 years to monitor the long-term safety of AGN-151597.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria.

1. Age >= 18 years.
2. Signed and dated written informed consent obtained from the patient.
3. Ability to comply with testing and all protocol tests.

Exclusion Criteria:

Any one of the following will exclude patients from being enrolled into the study:

1. Unable or unwilling to meet requirements of the study.
2. Participation in a clinical study (ocular or non-ocular) with an investigational drug, agent or therapy in the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - University of California San Francisco - Mission Bay /ID# 235717, San Francisco, California
  - Cincinnati Eye Institute- Edgewood /ID# 236713, Edgewood, Kentucky
  - Duke Eye Center /ID# 235715, Durham, North Carolina
  - Retina Foundation of the Southwest /ID# 235199, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Simunovic MP, Shen W, Lin JY, Protti DA, Lisowski L, Gillies MC. Optogenetic approaches to vision restoration. Exp Eye Res. 2019 Jan;178:15-26. doi: 10.1016/j.exer.2018.09.003. Epub 2018 Sep 13. PMID 30218651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 participants were enrolled in the study in the United States.
Pre-assignment Details: The Safety Population included all enrolled participants who received at least 1 dose of study treatment and was used for all analyses.
Groups:
- Phase 1: Low Dose: Three participants were enrolled and received the lowest dose of AGN-151597 (Low). After completion of the 2-year core study visits, participants could have enrolled in a long-term follow-up for an additional 3 years to monitor the long term safety of AGN-15197.
- Phase 1: Mid Dose: Four participants were enrolled and received a higher dose of AGN-151597 (Mid). After completion of the 2-year core study visits, participants could have enrolled in a long-term follow-up for an additional 3 years to monitor the long term safety of AGN-15197.
- Phase 1: High Dose: Three participants were enrolled and received the highest dose of AGN-151597 (High). After completion of the 2-year core study visits, participants could have enrolled in a long-term follow-up for an additional 3 years to monitor the long term safety of AGN-15197.
- Phase 2: High Dose: Four participants were enrolled in Phase 2a and received the highest dose of AGN-151597 (High) from Phase 1. After completion of the 2-year core study visits, participants could have enrolled in a long-term follow-up for an additional 3 years to monitor the long term safety of AGN-15197.
Period: Open Label Treatment Period
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Started | 3 | 4 | 3 | 4
Completed | 3 | 4 | 2 | 2
Not Completed | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Long-Term Follow-up
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Started | 1 (2 participants who completed Treatment Period did not enter the Long-Term Follow-up Period.) | 4 | 2 | 2
Completed | 0 | 4 | 2 | 1
Not Completed | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose | Total
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (17.09) | 58.8 (4.99) | 64.7 (8.33) | 50.0 (24.12) | 59.1 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 | 4
  Male | 2 | 2 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 3 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 1 | 4 | 3 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Grade 3 or Greater Adverse Event (AE) Considered Related to AGN-151597
Description: An adverse event is any untoward medical occurrence in a subject or clinical investigation patient administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Baseline (Day 1) to 6 Months
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 4
participants | 0 | 0 | 0 | 0

2. Primary Outcome: Visual Acuity in the Study Eye at Baseline and Month 6
Description: Visual acuity of the study eye (with fellow eye covered) was measured using low vision assessment of count fingers, hand motion, and light perception.
  For count fingers testing, the examiner's hand presenting 1, 2, or 5 fingers is held 2 feet in front of the eye being examined. If the participant correctly identifies three of five presentations, then count fingers vision is noted. If not, then the participant must be tested for hand motion vision.
  For hand motion testing, the examiner's hand is extended 2 feet in front of the eye and moved horizontally or vertically. If the participant correctly identifies hand movement four out of five times, then hand motion vision is noted. If not, then the participant is tested for light perception.
  For light perception testing, a beam of light is directed in and out of the eye at least four times from a distance of 3 feet. If the participant correctly perceives the light, vision should be recorded as yes to light perception.
Time Frame: Baseline (Day 1), 6 Months
Population: Safety Population. Number Analyzed is the number of participants who had the assessment for the parameter at the specified visit. Although subjects who passed the Count Fingers assessment did not need to be evaluated for the Hand Motion assessment, and subjects who passed the Hand Motion assessment did not need to be evaluated further for the Light Perception Assessment, some participants who passed the previous assessments were still evaluated in error for subsequent assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 4
Participants
  Count Fingers (Baseline) | 0 | 0 | 0 | 0
  Count Fingers (6 months): number analyzed (Participants) | 3 | 4 | 3 | 2
  Count Fingers (6 months) | 0 | 0 | 0 | 0
  Hand Motion (Baseline) | 0 | 0 | 1 | 1
  Hand Motion (6 months): number analyzed (Participants) | 3 | 4 | 3 | 2
  Hand Motion (6 months) | 0 | 1 | 1 | 1
  Light Perception (Baseline): number analyzed (Participants) | 3 | 4 | 2 | 4
  Light Perception (Baseline) | 3 | 4 | 1 | 4
  Light Perception (6 months): number analyzed (Participants) | 3 | 3 | 2 | 2
  Light Perception (6 months) | 3 | 3 | 1 | 2

3. Primary Outcome: Change From Baseline at Month 6 in Full Field Sensitivity in the Study Eye - Blue Light Threshold
Description: The light sensitivity of the visual field was measured by recording the threshold at which a participant reported seeing the dimmest flash. A negative value indicates an increase in sensitivity from baseline.
Time Frame: Baseline (Day 1) to Month 6
Population: Safety Population. The Overall Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and specified postbaseline visit (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: Decibels
Groups:
- Phase 1: Low Dose: Three participants were enrolled and received a low dose of AGN-151597 (Low). After completion of the 2-year core study visits, participants could have enrolled in a long-term follow-up for an additional 3 years to monitor the long term safety of AGN-15197.
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 1 | 2
Decibels |  | 0.404 (NA) — Not calculable for n=1 | -6.600 (NA) — Not calculable for n=1 | 1.235 (5.1760)

4. Primary Outcome: Change From Baseline at Month 6 in Full Field Sensitivity in the Study Eye - Red Light Threshold
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Month 6
Population: Safety Population. The Overall Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and at the 6-month visit (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 1 | 2
Decibels |  | 0.903 (NA) — Not calculable for n=1 | -10.900 (NA) — Not calculable for n=1 | -0.232 (1.2601)

5. Primary Outcome: Change From Baseline at Month 6 in Full Field Sensitivity in the Study Eye - White Light Threshold
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 2 | 1 | 2
Decibels | 0.109 (1.2459) | -6.572 (9.3734) | -4.700 (NA) — Not calculable for n=1 | -1.887 (2.0520)

6. Primary Outcome: Change From Baseline at Month 6 in Ambulation in the Study Eye (Time)
Description: Evaluated a participant's ability to navigate within a dark room. The time from the start to stop and the distance from the center of the lit panel to where the participant stopped or touched the target (panel) were recorded. The test was first performed binocularly, then on the study eye (with non-study eye patched). A negative value indicates a decrease from baseline in time or distance from start to stop (improvement).
Time Frame: Baseline (Day 1) to Month 6
Population: Safety Population. The Overall Number Analyzed is the number of participants who completed the assessment with evaluable data (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 4 | 2 | 2
seconds | -15.50 (20.506) | -7.25 (10.500) | -0.50 (0.707) | -4.50 (6.364)

7. Primary Outcome: Change From Baseline at Month 6 in Ambulation in the Study Eye (Distance)
Description: as for outcome 6
Time Frame: Baseline (Day 1) to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 4 | 2 | 2
meters | -0.45 (1.025) | 0.16 (0.649) | -0.27 (0.410) | 0.02 (0.028)

8. Primary Outcome: Intraocular Pressure (IOP) Measurements in the Study Eye
Description: Intraocular pressure was measured using the Goldmann applanation tonometer or a hand-held tonometer (same instrument used for each participant throughout the study, when possible). Measurements were taken at baseline (pre-injection) and at 6 months.
Time Frame: Baseline (Day 1), 6 Months
Population: Safety Population. Number Analyzed is the number of participants who had the assessment for the parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 4
mmHg
  Baseline (pre-injection) | 13.3 (0.58) | 13.5 (1.91) | 18.7 (3.51) | 14.0 (2.94)
  Month 6: number analyzed (Participants) | 3 | 3 | 3 | 2
  Month 6 | 13.3 (0.58) | 15.3 (5.03) | 17.0 (3.00) | 15.0 (4.24)

9. Primary Outcome: Anatomical Parameters as Measured in the Study Eye by Color Fundus Photography and Autofluorescence
Description: A standardized procedure for the collection of single, non-stereo images of the fundus of both eyes was obtained using the same equipment for each participant throughout the study.
  Evidence of increased inflammation, hemorrhage, retinal detachment, RPE disturbance or atrophy in the fovea, and any changes from baseline visit were documented. Any changes from baseline in fundus autofluorescence were also documented.
Time Frame: Baseline (Day 1), 6 Months
Population: Safety Population. The Number Analyzed is the number of participants who completed the assessment with evaluable data the specified visit (whose vision abilities allowed them to participate in the testing).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 4
Participants
  Any Evidence of Inflammation (Baseline): number analyzed (Participants) | 1 | 3 | 3 | 3
  Any Evidence of Inflammation (Baseline) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Hemorrhage (Baseline): number analyzed (Participants) | 1 | 3 | 3 | 3
  Any Evidence of Retinal Hemorrhage (Baseline) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Detachment (Baseline): number analyzed (Participants) | 1 | 3 | 3 | 3
  Any Evidence of Retinal Detachment (Baseline) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Baseline): number analyzed (Participants) | 1 | 3 | 3 | 3
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Baseline) | 1 | 2 | 2 | 3
  Any Evidence of Atrophy in the Fovea (Baseline): number analyzed (Participants) | 1 | 3 | 3 | 3
  Any Evidence of Atrophy in the Fovea (Baseline) | 1 | 2 | 1 | 1
  Any Evidence of Other findings (Baseline): number analyzed (Participants) | 1 | 3 | 3 | 3
  Any Evidence of Other findings (Baseline) | 0 | 0 | 1 | 1
  Any findings of Autofluorescence (Baseline): number analyzed (Participants) | 1 | 2 | 2 | 2
  Any findings of Autofluorescence (Baseline) | 1 | 2 | 2 | 2
  Any Evidence of Inflammation (Month 6): number analyzed (Participants) | 1 | 3 | 3 | 1
  Any Evidence of Inflammation (Month 6) | 0 | 0 | 0 | 1
  Any Evidence of Retinal Hemorrhage (Month 6): number analyzed (Participants) | 1 | 3 | 3 | 1
  Any Evidence of Retinal Hemorrhage (Month 6) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Detachment (Month 6): number analyzed (Participants) | 1 | 3 | 3 | 1
  Any Evidence of Retinal Detachment (Month 6) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Month 6): number analyzed (Participants) | 1 | 3 | 3 | 2
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Month 6) | 1 | 2 | 1 | 2
  Any Evidence of Atrophy in the Fovea (Month 6): number analyzed (Participants) | 1 | 3 | 3 | 1
  Any Evidence of Atrophy in the Fovea (Month 6) | 1 | 2 | 1 | 0
  Any Evidence of Other findings (Month 6): number analyzed (Participants) | 1 | 3 | 3 | 1
  Any Evidence of Other findings (Month 6) | 0 | 0 | 1 | 1
  Any findings of Autofluorescence (Month 6): number analyzed (Participants) | 0 | 0 | 0 | 0

10. Primary Outcome: Change From Baseline at Month 6 in the Anatomical Parameters in the Study Eye as Measured by Spectral Domain-Optical Coherence Tomography (SD-OCT) - Total Retinal Nerve Fibre Layer Volume
Description: Qualitative assessment of the change in retinal cross-sectional appearance in the study eye from Baseline at month 6 as Measured by SD-OCT.
Time Frame: Baseline (Day 1) to Month 6
Population: Safety Population. The Overall Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and the 6-month visit (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 2 | 0
mm3 |  | 1.760 (NA) — Not calculable for n=1 | 0.005 (0.0212) |

11. Primary Outcome: Change From Baseline at Month 6 in the Anatomical Parameters in the Study Eye as Measured by Spectral Domain-Optical Coherence Tomography (SD-OCT) - Total Ganglion Cell and Inner Plexiform Layer Volume
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 2 | 0
mm3 |  | 0.180 (NA) — Not calculable for n=1 | -0.055 (0.0636) |

12. Primary Outcome: Change From Baseline at Month 6 in the Anatomical Parameters in the Study Eye as Measured by Spectral Domain-Optical Coherence Tomography (SD-OCT) - Total Retinal Volume
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 0 | 2 | 0
mm3 |  |  | 0.570 (0.7495) |

13. Primary Outcome: Change From Baseline at Month 6 in the Anatomical Parameters in the Study Eye as Measured by Spectral Domain-Optical Coherence Tomography (SD-OCT) - Total Retinal Thickness
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 2 | 0
um |  | 14.0 (NA) — Not calculable for n=1 | 60.0 (86.27) |

14. Secondary Outcome: Visual Acuity in the Study Eye at Months 3, 12, and 24
Description: as for outcome 2
Time Frame: 3, 12, and 24 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Mid Dose: Three participants were enrolled and received a higher dose of AGN-151597 (Mid). After completion of the 2-year core study visits, participants could have enrolled in a long-term follow-up for an additional 3 years to monitor the long term safety of AGN-15197.
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 4
Participants
  Count Fingers (3 months) | 0 | 0 | 0 | 0
  Count Fingers (12 months) | 0 | 0 | 0 | 0
  Count Fingers (24 months) | 0 | 0 | 0 | 0
  Hand Motion (3 months) | 0 | 2 | 1 | 1
  Hand Motion (12 months): number analyzed (Participants) | 2 | 4 | 3 | 3
  Hand Motion (12 months) | 0 | 1 | 1 | 1
  Hand Motion (24 months): number analyzed (Participants) | 3 | 4 | 2 | 1
  Hand Motion (24 months) | 0 | 1 | 2 | 0
  Light Perception (3 months): number analyzed (Participants) | 3 | 2 | 2 | 4
  Light Perception (3 months) | 3 | 2 | 1 | 4
  Light Perception (12 months): number analyzed (Participants) | 2 | 3 | 2 | 3
  Light Perception (12 months) | 2 | 3 | 1 | 3
  Light Perception (24 months): number analyzed (Participants) | 3 | 3 | 0 | 1
  Light Perception (24 months) | 3 | 3 |  | 1

15. Secondary Outcome: Change From Baseline at Months 3, 12, and 24 in Full Field Sensitivity in the Study Eye - Blue Light Threshold
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Months 3, 12, and 24
Population: Safety Population. The Overall Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and at least one of the postbaseline visits (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 2 | 4
Decibels
  Blue Light Threshold (3 months) |  | -1.097 (NA) — Not calculable for n=1 | -10.050 (12.7986) | -0.475 (2.7628)
  Blue Light Threshold (12 months): number analyzed (Participants) | 0 | 1 | 2 | 3
  Blue Light Threshold (12 months) |  | 0.008 (NA) — Not calculable for n=1 | -7.300 (7.2125) | -0.905 (3.0047)
  Blue Light Threshold (24 months): number analyzed (Participants) | 0 | 1 | 1 | 1
  Blue Light Threshold (24 months) |  | 3.332 (NA) — Not calculable for n=1 | -8.100 (NA) — Not calculable for n=1 | -1.121 (NA) — Not calculable for n=1

16. Secondary Outcome: Change From Baseline at Months 3, 12, and 24 in Full Field Sensitivity in the Study Eye - Red Light Threshold
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Months 3, 12, and 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 2 | 2 | 4
Decibels
  Red Light Threshold (3 months) |  | 1.259 (1.9389) | -5.700 (8.7681) | -1.046 (1.9526)
  Red Light Threshold (12 months): number analyzed (Participants) | 0 | 1 | 2 | 3
  Red Light Threshold (12 months) |  | -0.301 (NA) — Not calculable for n=1 | -5.100 (8.3439) | 1.537 (4.5122)
  Red Light Threshold (24 months): number analyzed (Participants) | 0 | 2 | 1 | 1
  Red Light Threshold (24 months) |  | 2.901 (6.2119) | -10.000 (NA) — Not calculable for n=1 | -1.876 (NA) — Not calculable for n=1

17. Secondary Outcome: Change From Baseline at Months 3, 12, and 24 in Full Field Sensitivity in the Study Eye - White Light Threshold
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Months 3, 12, and 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
Decibels
  White Light Threshold (3 months) | -0.666 (6.6383) | -1.988 (2.1383) | -7.500 (11.7380) | -0.066 (2.4312)
  White Light Threshold (12 months): number analyzed (Participants) | 2 | 2 | 2 | 3
  White Light Threshold (12 months) | -0.351 (2.2642) | -4.414 (7.3348) | -9.500 (3.8184) | -1.699 (1.2484)
  White Light Threshold (24 months): number analyzed (Participants) | 2 | 2 | 1 | 1
  White Light Threshold (24 months) | 3.882 (1.5373) | -5.734 (12.5384) | -3.000 (NA) — Not calculable for n=1 | -3.887 (NA) — Not calculable for n=1

18. Secondary Outcome: Change From Baseline at Months 3, 12, and 24 in Ambulation Light-Guided Walking Test in the Study Eye (Time)
Description: as for outcome 6
Time Frame: Baseline (Day 1) to Months 3, 12, and 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 4 | 2 | 4
seconds
  Mean Time (seconds) (3 months) | -19.00 (14.142) | -6.00 (13.441) | 0.00 (0.000) | 1.50 (2.082)
  Mean Time (seconds) (12 months): number analyzed (Participants) | 2 | 4 | 2 | 3
  Mean Time (seconds) (12 months) | -15.50 (21.920) | -12.00 (16.573) | -3.00 (4.243) | 0.00 (4.000)
  Mean Time (seconds) (24 months): number analyzed (Participants) | 2 | 4 | 2 | 1
  Mean Time (seconds) (24 months) | -16.00 (25.456) | -11.50 (17.253) | -2.00 (1.414) | -6.00 (NA) — Not calculable for n=1

19. Secondary Outcome: Change From Baseline at Months 3, 12, and 24 in Ambulation Light-Guided Walking Test in the Study Eye (Distance)
Description: as for outcome 6
Time Frame: Baseline (Day 1) to Months 3, 12, and 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 4 | 2 | 3
meters
  Mean Distance (meters) (3 months) | -0.57 (1.011) | 0.07 (0.369) | -0.16 (0.247) | -0.01 (0.012)
  Mean Distance (meters) (12 months): number analyzed (Participants) | 2 | 4 | 2 | 2
  Mean Distance (meters) (12 months) | -0.26 (1.344) | 0.20 (0.529) | 0.38 (0.467) | 0.02 (0.000)
  Mean Distance (meters) (24 months): number analyzed (Participants) | 2 | 4 | 2 | 1
  Mean Distance (meters) (24 months) | 0.13 (0.884) | 0.14 (0.638) | -0.19 (0.318) | -0.02 (NA) — Not calculable for n=1

20. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Object Detection and Discrimination Scores
Description: Participants were to perform two tests concurrently, first identifying if a light displayed on an LED screen can be seen and then if a series of standard images (square, circle, triangle, or star) presented on the screen can be identified. The shapes were presented in blue or red at varying intensities. Data on light color and threshold intensity of the light was collected; shape detection data was not collected. The change from baseline in threshold intensity at 3, 6, and 24 months is reported. A negative change from baseline suggests an improvement.
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: cd/m2
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 0 | 1 | 2
cd/m2
  Blue Threshold Intensity (3 months) | -68.939 (146.2578) |  | 5.998 (NA) — Not calculable for n=1. | -1.865 (11.8409)
  Red Threshold Intensity (3 months): number analyzed (Participants) | 1 | 0 | 0 | 2
  Red Threshold Intensity (3 months) | -18925.624 (NA) — Not calculable for n=1. |  |  | 10323.422 (14244.9927)
  Blue Threshold Intensity (6 months) | -124.924 (184.2505) |  | 0.000 (NA) — Not calculable for n=1. | 0.515 (2.3009)
  Red Threshold Intensity (6 months): number analyzed (Participants) | 1 | 0 | 1 | 2
  Red Threshold Intensity (6 months) | -18952.831 (NA) — Not calculable for n=1. |  | -184.612 (NA) — Not calculable for n=1. | 3.195 (8.0718)
  Blue Threshold Intensity (24 months): number analyzed (Participants) | 1 | 0 | 0 | 1
  Blue Threshold Intensity (24 months) | 334.603 (NA) — Not calculable for n=1. |  |  | 199.747 (NA) — Not calculable for n=1.
  Red Threshold Intensity (24 months): number analyzed (Participants) | 0 | 0 | 0 | 1
  Red Threshold Intensity (24 months) |  |  |  | -1.266 (NA) — Not calculable for n=1.

21. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Visual Evoked Potential (VEP) Scores in the Study Eye (SE/0.974 Amplitude)
Description: Visual Evoked Potential (VEP) is an eye assessment that measures how the brain responds to visual stimuli. The pattern of visual evoked potentials was obtained from each eye using a VEP stimulator according to standard protocols. Three different visual stimuli were assessed. Amplitude measures how strong the signal is when your brain responds to visual stimuli. A higher amplitude indicates an improvement and a lower amplitude indicates a worsening outcome. Latency is the time it takes for the signal to reach the brain after the visual stimulus is presented. A shorter latency indicates an improvement from baseline; a longer latency indicates a worsening outcome.
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: Safety Population. The Overall Number of Participants Analyzed is the number of participants who completed assessment with evaluable data at baseline and at least one postbaseline visit at Month 3, Month 6, or Month 24. The Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and specified postbaseline visit (whose vision abilities allowed them to participate in the testing)
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 0 | 0 | 1
mV
  SE/0.974 Amplitude (mV) - 3 months: number analyzed (Participants) | 1 | 0 | 0 | 1
  SE/0.974 Amplitude (mV) - 3 months | 0.0 (NA) — Not calculable for n=1 |  |  | 1.0 (NA) — Not calculable for n=1
  SE/0.974 Amplitude (mV) - 6 months: number analyzed (Participants) | 0 | 0 | 0 | 0
  SE/0.974 Amplitude (mV) - 24 months: number analyzed (Participants) | 1 | 0 | 0 | 0
  SE/0.974 Amplitude (mV) - 24 months | 47.0 (NA) — Not calculable for n=1 |  |  |

22. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Visual Evoked Potential (VEP) Scores in the Study Eye (SE/0.649 Amplitude)
Description: as for outcome 21
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: Safety Population. The Overall Number of Participants Analyzed is the number of participants assessed at baseline. The Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and specified postbaseline visit (whose vision abilities allowed them to participate in the testing)
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 0 | 0 | 1
mV
  SE/0.649 Amplitude (mV) - 3 months: number analyzed (Participants) | 1 | 0 | 0 | 1
  SE/0.649 Amplitude (mV) - 3 months | 0.0 (NA) — Not calculable for n=1 |  |  | 0.0 (NA) — Not calculable for n=1
  SE/0.649 Amplitude (mV) - 6 months: number analyzed (Participants) | 0 | 0 | 0 | 0
  SE/0.649 Amplitude (mV) - 24 months: number analyzed (Participants) | 3 | 0 | 0 | 0
  SE/0.649 Amplitude (mV) - 24 months | 10.3 (19.66) |  |  |

23. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Visual Evoked Potential (VEP) Scores in the Study Eye (SE/0.216 Amplitude)
Description: as for outcome 21
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 0 | 0 | 1
mV
  SE/0.216 Amplitude (mV) - 3 months: number analyzed (Participants) | 1 | 0 | 0 | 1
  SE/0.216 Amplitude (mV) - 3 months | -4.0 (NA) — Not calculable for n=1 |  |  | 0.0 (NA) — Not calculable for n=1
  SE/0.216 Amplitude (mV) - 6 months: number analyzed (Participants) | 0 | 0 | 0 | 0
  SE/0.216 Amplitude (mV) - 24 months: number analyzed (Participants) | 2 | 0 | 0 | 0
  SE/0.216 Amplitude (mV) - 24 months | 40.5 (55.86) |  |  |

24. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Visual Evoked Potential (VEP) Scores in the Study Eye (SE/0.974 Latency)
Description: as for outcome 21
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 2 | 0 | 1 | 1
msec
  SE/0.974 Latency (msec) - 3 months: number analyzed (Participants) | 1 | 0 | 0 | 1
  SE/0.974 Latency (msec) - 3 months | -1.0 (NA) — Not calculable for n=1 |  |  | 25.0 (NA) — Not calculable for n=1
  SE/0.974 Latency (msec) - 6 months: number analyzed (Participants) | 0 | 0 | 0 | 0
  SE/0.974 Latency (msec) - 24 months: number analyzed (Participants) | 1 | 0 | 0 | 0
  SE/0.974 Latency (msec) - 24 months | 40.0 (NA) — Not calculable for n=1 |  |  |

25. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Visual Evoked Potential (VEP) Scores in the Study Eye (SE/0.649 Latency)
Description: as for outcome 21
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 0 | 0 | 1
msec
  SE/0.649 Latency (msec) - 3 months: number analyzed (Participants) | 1 | 0 | 0 | 1
  SE/0.649 Latency (msec) - 3 months | 13.0 (NA) — Not calculable for n=1 |  |  | 15.0 (NA) — Not calculable for n=1
  SE/0.649 Latency (msec) - 6 months: number analyzed (Participants) | 0 | 0 | 0 | 0
  SE/0.649 Latency (msec) - 24 months: number analyzed (Participants) | 3 | 0 | 0 | 0
  SE/0.649 Latency (msec) - 24 months | -6.3 (10.02) |  |  |

26. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Visual Evoked Potential (VEP) Scores in the Study Eye (SE/0.216 Latency)
Description: as for outcome 21
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 0 | 0 | 1
msec
  SE/0.216 Latency (msec) - 3 months: number analyzed (Participants) | 1 | 0 | 0 | 1
  SE/0.216 Latency (msec) - 3 months | -21.0 (NA) — Not calculable for n=1 |  |  | 7.0 (NA) — Not calculable for n=1
  SE/0.216 Latency (msec) - 6 months: number analyzed (Participants) | 0 | 0 | 0 | 0
  SE/0.216 Latency (msec) - 24 months: number analyzed (Participants) | 2 | 0 | 0 | 0
  SE/0.216 Latency (msec) - 24 months | 22.0 (5.66) |  |  |

27. Secondary Outcome: Change From Baseline at Months 6 and 24 in Electroretinogram (ERG) Scores in the Study Eye (Amplitude)
Description: Full field electroretinography based on standards set by the ERG Standardization Committee of the International Society for Clinical Electrophysiology of Vision (ISCEV) was performed at the Screening visit, 6 months, and at 24 months. ERG tests how well the light sensitive part of the eye (retina) is working. Several assessments were performed to evaluate how well different parts of the retina respond to light in different settings. Amplitude is the strength of the electrical signal that the retina produces in response to light during an ERG test. Higher amplitude in A-wave or b-wave indicates improvement; lower amplitude indicates worsening.
Time Frame: Baseline (Day 1) to Months 6 and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 3
uV
  Dark Adapted 0.01 ERG b-wave (uV) - 6 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Dark Adapted 0.01 ERG b-wave (uV) - 6 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Dark Adapted 3 ERG a-wave (uV) - 6 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Dark Adapted 3 ERG a-wave (uV) - 6 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Dark Adapted 3 ERG b-wave (uV) - 6 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Dark Adapted 3 ERG b-wave (uV) - 6 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 ERG a-wave (uV) - 6 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Light Adapted 3 ERG a-wave (uV) - 6 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 ERG b-wave (uV) - 6 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Light Adapted 3 ERG b-wave (uV) - 6 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Light Adapted 30 Flicker Amplitude (uV) - 6 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Light Adapted 30 Flicker Amplitude (uV) - 6 months | -0.0423 (0.14301) | -0.2318 (0.28927) | 0.0000 (0.0000) | 0.0000 (NA) — Not calculable for n=1
  Dark Adapted 0.01 ERG b-wave (uV) - 24 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Dark Adapted 0.01 ERG b-wave (uV) - 24 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Dark Adapted 3 ERG a-wave (uV) - 24 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Dark Adapted 3 ERG a-wave (uV) - 24 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Dark Adapted 3 ERG b-wave (uV) - 24 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Dark Adapted 3 ERG b-wave (uV) - 24 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 ERG a-wave (uV) - 24 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Light Adapted 3 ERG a-wave (uV) - 24 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 ERG b-wave (uV) - 24 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Light Adapted 3 ERG b-wave (uV) - 24 months | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (NA) — Not calculable for n=1
  Light Adapted 30 Flicker Amplitude (uV) - 24 months: number analyzed (Participants) | 3 | 4 | 2 | 1
  Light Adapted 30 Flicker Amplitude (uV) - 24 months | 0.7897 (0.95459) | -0.2630 (0.26256) | 0.0000 (0.0000) | 0.0000 (NA) — Not calculable for n=1

28. Secondary Outcome: Change From Baseline at Months 6 and 24 in Electroretinogram (ERG) Scores in the Study Eye (Latency)
Description: Full field electroretinography based on standards set by the ERG Standardization Committee of the International Society for Clinical Electrophysiology of Vision (ISCEV) was performed at the Screening visit, 6 months, and at 24 months. ERG tests how well the light sensitive part of the eye (retina) is working. Several assessments were performed to evaluate how well different parts of the retina respond to light in different settings. Amplitude is the strength of the electrical signal that the retina produces in response to light during an ERG test. Latency is the time it takes for the retina to respond after a light is flashed in the eye during an ERG test. Shorter latency indicates an improvement; longer latency indicates a worsening.
Time Frame: Baseline (Day 1) to Months 6 and 24
Population: Safety Population. The Overall Number of Participants Analyzed is the number of participants who completed assessment with evaluable data at baseline and at least one postbaseline visit at Month 6 or Month 24. The Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and specified postbaseline visit (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 3 | 0 | 3
msec
  Dark Adapted 0.01 ERG Latency (msec) - 6 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Dark Adapted 0.01 ERG Latency (msec) - 6 months | 0.0 (0.0) | 0.0 (0.0) |  | 0.0 (NA) — Not calculable for n=1
  Dark Adapted 3 ERG Latency (msec) - 6 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Dark Adapted 3 ERG Latency (msec) - 6 months | 0.0 (0.0) | 0.0 (0.0) |  | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 ERG Latency (msec) - 6 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Light Adapted 3 ERG Latency (msec) - 6 months | 0.0 (0.0) | 0.0 (0.0) |  | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 Flicker Latency (msec) - 6 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Light Adapted 3 Flicker Latency (msec) - 6 months | -20.0 (22.54) | -24.3 (37.07) |  | 0.0 (NA) — Not calculable for n=1
  Dark Adapted 0.01 ERG Latency (msec) - 24 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Dark Adapted 0.01 ERG Latency (msec) - 24 months | 0.0 (0.0) | 0.0 (0.0) |  | 0.0 (NA) — Not calculable for n=1
  Dark Adapted 3 ERG Latency (msec) - 24 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Dark Adapted 3 ERG Latency (msec) - 24 months | 0.0 (0.0) | 0.0 (0.0) |  | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 ERG Latency (msec) - 24 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Light Adapted 3 ERG Latency (msec) - 24 months | 0.0 (0.0) | 0.0 (0.0) |  | 0.0 (NA) — Not calculable for n=1
  Light Adapted 3 Flicker Latency (msec) - 24 months: number analyzed (Participants) | 3 | 3 | 0 | 1
  Light Adapted 3 Flicker Latency (msec) - 24 months | -4.7 (23.16) | -40.3 (17.39) |  | 0.0 (NA) — Not calculable for n=1

29. Secondary Outcome: Change From Baseline at Months 3, 6, and 24 in Composite Score of National Eye Institute (NEI) Visual Functioning Questionnaire (VFQ-25) Scores
Description: Change in quality of life, based on composite scores of the NEI VFQ-25 from Baseline at 3, 6, and 24 months. The NEI VFQ-25 consists of 25 vision-targeted questions that represent 11 vision-related quality of life subscales and one general health item. The 11 subscales are general vision, difficulty with near vision activities, difficulty with distance vision activities, limitation in social functioning due to vision, role limitation due to vision, dependency on others due to vision, mental health symptoms due to vision, driving difficulties, limitation with peripheral vision, limitation with color vision, and ocular pain. NEI VFQ-25 scores range from 0 to 100, with a higher score representing better functioning. A positive value change from baseline indicates an improvement in vision-related quality of life.
Time Frame: Baseline (Day 1) to Months 3, 6, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 4
score on a scale
  Month 3 | 4.3 (9.65) | 5.5 (6.18) | -5.3 (0.84) | 0.9 (14.76)
  Month 6: number analyzed (Participants) | 3 | 4 | 3 | 2
  Month 6 | 4.8 (14.37) | 6.2 (7.45) | -6.6 (3.37) | 9.4 (18.27)
  Month 24: number analyzed (Participants) | 3 | 4 | 2 | 1
  Month 24 | 8.3 (9.48) | 3.0 (6.86) | -7.4 (3.68) | 3.1 (NA) — Not calculable for n=1.

30. Secondary Outcome: Anatomical Parameters as Measured in the Study Eye by Color Fundus Photography and Autofluorescence
Description: A standardized procedure was used for the collection of single, non-stereo images of the fundus of both eyes using the same equipment for each participant throughout the study.
  Evidence of increased inflammation, hemorrhage, retinal detachment, RPE disturbance or atrophy in the fovea, and any changes from baseline visit were documented. Presence or absence of changes from baseline in fundus autofluorescence were also documented.
Time Frame: Months 3 and 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 3 | 4 | 3 | 4
Participants
  Any Evidence of Inflammation (Month 3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Any Evidence of Inflammation (Month 3) | 0 | 0 | 0 | 1
  Any Evidence of Retinal Hemorrhage (Month 3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Any Evidence of Retinal Hemorrhage (Month 3) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Detachment (Month 3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Any Evidence of Retinal Detachment (Month 3) | 0 | 0 | 0 | 0
  Any Evidence of Atrophy in the Fovea (Month 3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Any Evidence of Atrophy in the Fovea (Month 3) | 2 | 1 | 1 | 1
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Month 3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Month 3) | 2 | 1 | 1 | 2
  Any Findings of Autofluorescence (Month 3): number analyzed (Participants) | 0 | 0 | 0 | 0
  Any Findings of Autofluorescence (Month 3) | 0 | 0 | 0 | 0
  Any Evidence of Other findings (Month 3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Any Evidence of Other findings (Month 3) | 0 | 0 | 1 | 2
  Any Evidence of Inflammation (Month 24): number analyzed (Participants) | 3 | 3 | 2 | 1
  Any Evidence of Inflammation (Month 24) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Hemorrhage (Month 24): number analyzed (Participants) | 3 | 3 | 2 | 1
  Any Evidence of Retinal Hemorrhage (Month 24) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Detachment (Month 24): number analyzed (Participants) | 3 | 3 | 2 | 1
  Any Evidence of Retinal Detachment (Month 24) | 0 | 0 | 0 | 0
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Month 24): number analyzed (Participants) | 3 | 3 | 2 | 1
  Any Evidence of Retinal Pigment Epithelium (RPE) Disturbance (Month 24) | 3 | 2 | 1 | 1
  Any Evidence of Atrophy in the Fovea (Month 24): number analyzed (Participants) | 3 | 3 | 2 | 1
  Any Evidence of Atrophy in the Fovea (Month 24) | 3 | 2 | 0 | 0
  Any Evidence of Other findings (Month 24): number analyzed (Participants) | 3 | 3 | 2 | 1
  Any Evidence of Other findings (Month 24) | 0 | 0 | 0 | 0
  Any Findings of Autofluorescence (Month 24): number analyzed (Participants) | 0 | 0 | 0 | 0
  Any Findings of Autofluorescence (Month 24) | 0 | 0 | 0 | 0

31. Secondary Outcome: Change From Baseline at Months 3, 12, and 24 in the Anatomical Parameters in the Study Eye as Measured by Spectral Domain-OCT (SD-OCT) - Volume
Description: Qualitative assessment of the change in retinal cross-sectional appearance in the study eye from Baseline at Months 3, 12, and 24 as Measured by Spectral Domain-OCT (SD-OCT).
Time Frame: Baseline to Months 3, 12, and 24
Population: Safety Population. The Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and specified postbaseline visit (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 2 | 0
mm3
  Total Retinal Nerve Fibre Layer Volume (mm3) (3 months) |  | 0.350 (NA) — Not calculable for n=1 | 0.060 (0.1131) |
  Total Ganglion Cell and Inner Plexiform Layer Volume (mm3) (3 months) |  | 0.210 (NA) — Not calculable for n=1 | 0.070 (0.0990) |
  Total Retinal Volume (mm3) (3 months): number analyzed (Participants) | 0 | 0 | 2 | 0
  Total Retinal Volume (mm3) (3 months) |  |  | 0.945 (1.1809) |
  Total Retinal Nerve Fibre Layer Volume (mm3) (12 months) |  | -0.040 (NA) — Not calculable for n=1 | 0.080 (0.0212) |
  Total Ganglion Cell and Inner Plexiform Layer Volume (mm3) (12 months) |  | 0.050 (NA) — Not calculable for n=1 | 0.005 (0.2051) |
  Total Retinal Volume (mm3) (12 months): number analyzed (Participants) | 0 | 0 | 2 | 0
  Total Retinal Volume (mm3) (12 months) |  |  | 0.085 (0.0919) |
  Total Retinal Nerve Fibre Layer Volume (mm3) (24 months) |  | -0.060 (NA) — Not calculable for n=1 | 0.060 (0.1131) |
  Total Ganglion Cell and Inner Plexiform Layer Volume (mm3) (24 months) |  | 0.210 (NA) — Not calculable for n=1 | -0.065 (0.1202) |
  Total Retinal Volume (mm3) (24 months): number analyzed (Participants) | 0 | 0 | 2 | 0
  Total Retinal Volume (mm3) (24 months) |  |  | 0.135 (0.6152) |

32. Secondary Outcome: Change From Baseline at Months 3, 12, and 24 in the Anatomical Parameters in the Study Eye as Measured by Spectral Domain-OCT (SD-OCT) - Total Retinal Thickness
Description: as for outcome 31
Time Frame: Baseline to Months 3, 12, and 24
Population: Safety Population. The Overall Number Analyzed is the number of participants who completed the assessment with evaluable data at both baseline and the specified postbaseline visit (whose vision abilities allowed them to participate in the testing).
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
Number analyzed (Participants) | 0 | 1 | 2 | 0
um
  Total Retinal Thickness (um) (3 months) |  | 29.0 (NA) — Not calculable for n=1 | 63.0 (83.44) |
  Total Retinal Thickness (um) (12 months) |  | 12.0 (NA) — Not calculable for n=1 | 9.5 (12.02) |
  Total Retinal Thickness (um) (24 months) |  | 17.0 (NA) — Not calculable for n=1 | -1.0 (8.49) |

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from time of informed consent to the end of the study. The median time participants were followed was 885.0 days for Phase 1 (low dose); 1991.5 days for Phase 1 (mid dose); 1814.0 days for Phase 1 (high dose); and 800.5 days for Phase 2 (high dose).
Arm/Group | Phase 1: Low Dose | Phase 1: Mid Dose | Phase 1: High Dose | Phase 2: High Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 2/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Low Dose (N=3) | Phase 1: Mid Dose (N=4) | Phase 1: High Dose (N=3) | Phase 2: High Dose (N=4)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Low Dose (N=3) | Phase 1: Mid Dose (N=4) | Phase 1: High Dose (N=3) | Phase 2: High Dose (N=4)
ANTERIOR CHAMBER CELL (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLEPHARITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CATARACT NUCLEAR (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CATARACT SUBCAPSULAR (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
IRITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OCULAR HYPERTENSION (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VITREAL CELLS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VITREOUS DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
VITRITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SWELLING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FUNGAL FOOT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SIALOADENITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BENIGN NEOPLASM OF EYELID (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02556736/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02556736/SAP_003.pdf